CLINICAL TRIAL: NCT07008560
Title: Evaluation of Spatiotemporal Associations Between the COVID-19 Pandemic and the Incidence of Cancer Diagnoses in Bavaria, Germany: A Registry-based Study (PanSCan)
Brief Title: Spatiotemporal Associations Between the COVID-19 Pandemic and Cancer Diagnoses in Bavaria
Acronym: PanSCan
Status: Active, not recruiting | Type: Observational
Sponsor: Bavarian Cancer Registry (Other Government)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-1014
Record Dates: First submitted 2025-05-21; First posted 2025-06-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Cancer registration; Registry data; Population-based analysis; Incidence; COVID-19; Pandemics; Cancer
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bavarian Cancer Registry Cohort (2018-2023): The study cohort consists of all incident cancer cases diagnosed in individuals aged 18 years and older in Bavaria, Germany, between January 1, 2018, and December 31, 2023. Eligible cases were identified through the Bavarian Cancer Registry and include carcinoma in situ.

SUMMARY:
The COVID-19 pandemic has placed a significant strain on healthcare systems worldwide and has also impacted the diagnosis and treatment of cancer. In Germany, there was a notable decline in cancer diagnoses during the pandemic, partly due to delays in early detection and limited access to medical treatments.

This study examines how the number of cancer cases in Bavaria changed before and during the pandemic, taking various factors into account, such as the socioeconomic status of different regions, the age of affected individuals, and the severity of the pandemic in each region.

We aim to determine whether certain regions or specific types of tumors experienced greater declines in diagnoses, particularly for cancers with regular screening programs. The study seeks to provide a better understanding of how different social and geographical conditions influenced cancer diagnoses during the pandemic. These insights could help improve future preparedness for health crises like the pandemic and ensure that cancer treatment continues to function effectively even in times of crisis.

DETAILED DESCRIPTION:
The COVID-19 pandemic has exerted significant pressure on healthcare systems worldwide, particularly impacting the diagnosis and treatment of non-communicable diseases such as cancer. In Germany, substantial declines in cancer diagnoses have been observed, primarily due to delays in early detection and limited access to medical services during the pandemic. This study aims to investigate the regional and temporal variations in cancer incidence in Bavaria before and during the pandemic, taking into account socio-economic, demographic factors, and the severity of the pandemic.

This registry-based study utilizes data from the Bavarian Cancer Registry spanning from 2018 to 2023. The analysis adopts a spatiotemporal approach to examine changes in cancer incidence over time at the district level in Bavaria. A Bayesian spatiotemporal Poisson model with a Conditional Autoregressive (CAR) structure will be employed to account for both spatial and temporal variations, as well as spatial correlations between neighboring districts. The analysis will incorporate demographic characteristics, socio-economic status, tumor-specific data, and regional variations in the severity of the pandemic.

It is hypothesized that the pandemic has led to regional disparities in cancer incidence, with socio-economically disadvantaged areas potentially being more severely affected. Tumors associated with established screening programs, such as breast, colon, and cervical cancer, may have experienced a greater reduction in diagnoses compared to other cancer types.

The findings of this study will provide valuable insights into how geographical and socio-economic factors influenced cancer incidence during the pandemic and how these inequalities were exacerbated. The results could inform future health policies aimed at ensuring the continued accessibility of cancer detection and treatment, even during public health crises.

ELIGIBILITY:
Inclusion Criteria:

* All incident cancer cases among individuals aged 18 years and older, including carcinoma in situ, diagnosed between 2018 and 2023 within Bavaria and recorded in the Bavarian Cancer Registry.

Exclusion Criteria:

* Death Certificate Only (DCO) cases. as they lack essential clinical information and the recorded date of diagnosis is in most cases the date of death, leading to temporal distortions in incidence estimates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes all individuals aged 18 years and older with an incident diagnosis of cancer, including carcinoma in situ, recorded in the Bavarian Cancer Registry between 2018 and 2023.
Sampling Method: Non-Probability Sample
Enrollment: 438000 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Newly diagnosed cancer cases | 2018 to 2023
  Number of incident cancer cases per district and month in Bavaria, Germany

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Müller-Nordhorn, Prof. Dr., Principal Investigator — Bavarian Cancer Registry, Bavarian Health and Food Safety Authority
Locations (1):
- Bavarian Cancer Registry, Bavarian Health and Food Safety Authority, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Sharing of individual participant data (IPD) is not possible because the data originate from the Bavarian Cancer Registry, where legal restrictions and strict data protection regulations prohibit the disclosure of patient-level data. These measures are in place to safeguard participant privacy and ensure compliance with applicable ethical and legal standards.

REFERENCES:
- See also: Bavarian Cancer Registry — https://www.lgl.bayern.de/gesundheit/krebsregister/index_e.htm

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT07008560/SAP_000.pdf